CLINICAL TRIAL: NCT02936869
Title: Incentives for Postnatal Care Demand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Adanna Chukwuma, Doctoral Candidate, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HU-052
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Maternal Death; Neonatal Death
MeSH Terms: conditions — Maternal Death; Perinatal Death

ARMS (2):
- Control arm (No Intervention): Traditional birth attendants will receive an offer of two-weekly payouts per reported delivery they take that is verified by client.
- Referral incentive arm (Experimental): Traditional birth attendants will receive an offer of two-weekly payouts per reported delivery they take that is verified by client.
  Traditional birth attendants randomized to this arm will also receive an offer of two-weekly payouts per successful referral of delivery clients to postnatal care within 48 hours of delivery in a facility if verified.
  Interventions: Behavioral: Performance-based monetary incentives

INTERVENTIONS:
Behavioral: Performance-based monetary incentives
  Arms: Referral incentive arm

SUMMARY:
The purpose of this study is to identify the causal impact of performance-based monetary incentives in increasing postnatal care (PNC) referrals by traditional birth attendants (TBAs), via a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* community-based providers of antenatal and/or delivery care, and who are non-formally trained
* must be resident within the community
* must not plan to relocate over the intervention duration
* identified in partnership with community leadership
* be willing to participate fully in the study, including having their clients contacted for verification

Exclusion Criteria:

* plan to relocate over the intervention duration
* refusal to provide informed consent for the entire study protocol including agreeing to have their delivery clients contacted for verification

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adanna Chukwuma, MBBS, MSc., Principal Investigator — Harvard School of Public Health (HSPH); Margaret McConnell, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Jessica Cohen, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Chinyere Mbachu, MBBS, MPH, Principal Investigator — Health Policy Research Group

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for this study including all the variables used for the analysis are available for download on the Harvard Dataverse.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data on the Harvard Dataverse are available indefinitely as long as the website continues to host datasets.
Access Criteria: The data can be freely downloaded without permission.

REFERENCES:
- [Background] Itina SM. Characteristics of traditional birth attendants and their beliefs and practices in the Offot Clan, Nigeria. Bull World Health Organ. 1997;75(6):563-7. PMID 9509629
- [Background] Sibley LM, Sipe TA, Barry D. Traditional birth attendant training for improving health behaviours and pregnancy outcomes. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD005460. doi: 10.1002/14651858.CD005460.pub3. PMID 22895949
- [Background] Oyebola, B. C., Muhammad, F., Otunomeruke, A., & Galadima, A. (2014). Effect of Performance-Based Incentives for Traditional Birth Attendants on Access to Maternal and Newborn Health-care Facilities in Gombe State, Nigeria: A Pilot Study. Meeting Abstract. Lancet.
- [Background] WHO. (2004). Making Pregnancy Safer: The Critical Role of the Skilled Attendant - A Joint Statement by WHO, ICM, and FIGO. Geneva: World Health Organization.
- [Derived] Chukwuma A, Mbachu C, McConnell M, Bossert TJ, Cohen J. The impact of monetary incentives on referrals by traditional birth attendants for postnatal care in Nigeria. BMC Pregnancy Childbirth. 2019 May 20;19(1):150. doi: 10.1186/s12884-019-2313-8. PMID 31104629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community within 128 wards in Ebonyi State in August 2016.
Pre-assignment Details: Of the 269 TBAs identified through community leaders and facility heads that met the inclusion criteria and were recruited, 20 declined to participate and 27 could not be located at the given addresses.
Groups:
- Referral Incentive Arm: Traditional birth attendants will receive an offer of two-weekly payouts per reported delivery they take that is verified by client.
  Traditional birth attendants randomized to this arm will also receive an offer of two-weekly payouts per successful referral of delivery clients to postnatal care within 48 hours of delivery in a facility if verified.
  Performance-based monetary incentives
Period: Overall Study
Arm/Group | Control Arm | Referral Incentive Arm
Started | 104 | 103
Completed | 102 | 98
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 1 | 3
Not completed — Death | 0 | 1
Not completed — Legal Case | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Referral Incentive Arm | Total
Number analyzed (Participants) | 104 | 103 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.42308 (19.67241) | 44.75728 (16.23206) | 48.10628 (18.30641)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 97 | 198
  Male | 3 | 6 | 9
Number of participants lacking formal education [Number; unit: Participants] | 47 | 40 | 87
Average income per pregnancy [Mean (Standard Deviation); unit: Naira] | 1790.962 (1852.523) | 2265.437 (2992.071) | 2027.053 (2491.036)
Number of participants offering postnatal care [Number; unit: Participants] | 70 | 60 | 130
Monthly average of delivery clients [Mean (Standard Deviation); unit: clients] | 13.80769 (97.70553) | 9.553398 (48.90622) | 11.69082 (77.21418)
Number of participants that are literate in English [Number; unit: Participants] | 44 | 47 | 91
Number of participants that are literate in non-English Language [Number; unit: Participants] | 26 | 29 | 55
Number of participants who are leaders of any association [Number; unit: Participants] | 30 | 46 | 76
Number of participants who are members of any association [Number; unit: Participants] | 88 | 89 | 177
Number of participants who are the main income earner in household [Number; unit: Participants] | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Maternal Postnatal Care Referral
Description: The proportion of delivery clients that are successfully referred by the traditional birth attendant for postnatal care within 48 hours of delivery. For each delivery client that the traditional birth attendant reported, we visited at least three days after delivery to ascertain if they had been asked to visit the postnatal clinic, clarify if they had visited the clinic within 48 hours of delivery, and what care they had received (if yes). The team visited traditional birth attendants every two weeks to identify new clients. Where a new client was not up to three days post-delivery, the interview was postponed until the next visit by the team to the community. This occurred repeatedly, over a five-month frame.
Time Frame: Within 48 hours of delivery
Population: The analysis did not include information from the 7 TBAs lost to follow-up.
Measure: Number (95% Confidence Interval); unit: proportion of maternal clients referred
Arm/Group | Control Arm | Referral Incentive Arm
Number analyzed (Participants) | 102 | 98
proportion of maternal clients referred | 0.044 [-0.009 to 0.097] | 0.154 [0.079 to 0.229]

2. Secondary Outcome: Neonatal Postnatal Care Referral
Description: Proportion of neonates delivered by the traditional birth attendant that are successfully referred for postnatal care within 48 hours of delivery
Time Frame: Within 48 hours of delivery
Population: The analysis did not include data from 7 TBAs lost to follow-up.
Measure: Number (95% Confidence Interval); unit: proportion of neonates referred
Groups:
- Referral Incentive Arm: Traditional birth attendants will receive an offer of two-weekly payouts per reported delivery they take that is verified by client.
  Traditional birth attendants randomized to this arm will also receive an offer of two-weekly payouts per successful referral of maternal delivery clients to postnatal care within 48 hours of delivery in a facility if verified.
  Performance-based monetary incentives
Arm/Group | Control Arm | Referral Incentive Arm
Number analyzed (Participants) | 102 | 98
proportion of neonates referred | 0.032 [-0.015 to 0.079] | 0.126 [0.059 to 0.193]

ADVERSE EVENTS:
Time Frame: 5 months
Description: At recruitment, participants were informed about potential adverse events in a consent form. During follow-up, enumerators were required to ask for these and other events. All reportable events were to be forwarded to the Harvard Longwood Medical Area Institutional Review Board within 5 days of the PI becoming aware of the situation as per the Office of Human Research Administration policy.
Arm/Group | Control Arm | Referral Incentive Arm
All-Cause Mortality (participants affected / at risk) | 0/104 | 1/103
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/103
Other Adverse Events (participants affected / at risk) | 0/104 | 0/103

LIMITATIONS AND CAVEATS:
This study was concluded prior to schedule due to community conflict affecting the length of follow-up time; we relied on self-reports due to the poor information systems within the study context.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT02936869/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT02936869/SAP_001.pdf